CLINICAL TRIAL: NCT02546128
Title: LEICSTES = LEICeSter Tendon Extracorporeal Shockwave Studies Assessing the Benefits of the Addition of Extra-Corporeal Shockwave Treatment to a Structured Home-rehabilitation Programme for Patients With Tendinopathy.
Brief Title: LEICeSter Tendon Extracorporeal Shockwave Studies
Acronym: LEICSTES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UHL - 11401
Record Dates: First submitted 2015-06-15; First posted 2015-09-10 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2023-11

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): rehabilitation + "active-dose" ESWT (extra-corporeal shockwave therapy)
  Interventions: Device: Extra-Corporeal Shockwave Therapy (ESWT); Other: structured rehabilitation programme
- control (Placebo Comparator): rehabilitation + "placebo-dose" ESWT (extra-corporeal shockwave therapy)
  Interventions: Other: structured rehabilitation programme

INTERVENTIONS:
Device: Extra-Corporeal Shockwave Therapy (ESWT) — The use of ESWT from a commercially available machine at approved settings already in routine clinical use
  Arms: intervention
Other: structured rehabilitation programme — a structured and standardised rehabilitation programme specific to the tendon in question - already in routine clinical use

SUMMARY:
To assess whether the addition of Extra-corporeal Shockwave Therapy (ESWT) to a structured home-exercise programme has any additional benefit to patients with tendinopathies

DETAILED DESCRIPTION:
This involves patients with one of 6 different defined chronic tendinopathies. These individual sites are run as discrete sub-studies, with randomisation n occurring within sub-study grouping

ELIGIBILITY:
Inclusion Criteria:

1. Patients age >18
2. Symptoms (typically pain / stiffness) of at least 12 weeks of one of the following sites / conditions:

   1. Plantar fasciitis
   2. Insertional Achilles tendinopathy
   3. Mid-substance Achilles tendinopathy
   4. Patella tendinopathy
   5. Trochanteric pain syndrome (gluteus medius insertional tendinopathy / trochanteric bursitis)
   6. Tennis elbow
3. Referred for ESWT (shockwave) within the Sports Medicine Department
4. Objective imaging of tendon / structure confirming diagnosis and excluding tear or other structural injury (US or MRI acceptable)

Exclusion Criteria:

1. Patients with the normal exclusions for ESWT - including pre-existing skin injury over tendon site, recent steroid injection (within 6 weeks of ESWT starting), patients on anticoagulation, patients with haemophilia or other bleeding tendency, patients with current febrile illness
2. Previous ESWT treatment for the same condition

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
improvement in pain as assessed by a 0-10 visual analogue scale (VAS) | primary outcome 3 months

SECONDARY OUTCOMES:
improvement in pain as assessed by a 0-10 visual analogue scale (VAS) | secondary outcome at 6 months post treatment
improvement in function as assessed by several validated patient-rated outcome measures | 3 months and 6 months
  These will use validated patient-rated outcome measures (PROMS) already in routine use in this clinical service. This include specific site questions, for example patella tendon (VISA-P), achilles tendon (VISA-A), trochanteric pain (Oxford Hip Score, Non-Arthritic Hip Score), plantar fascia (revised foot function index, MOXFQ) all of which give a wider picture of the outcome of specific conditions. these are all fully detailed in the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wheeler, Principal Investigator — UHL NHS Trust
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

REFERENCES:
- [Derived] Wheeler PC, Dudson C, Calver R, Goodall D, Gregory KM, Singh H, Boyd KT. Three Sessions of Radial Extracorporeal Shockwave Therapy Gives No Additional Benefit Over "Minimal-Dose" Radial Extracorporeal Shockwave Therapy for Patients With Chronic Greater Trochanteric Pain Syndrome: A Double-Blinded, Randomized, Controlled Trial. Clin J Sport Med. 2022 Jan 1;32(1):e7-e18. doi: 10.1097/JSM.0000000000000880. PMID 33512943